CLINICAL TRIAL: NCT06533748
Title: SJALL23H: Combination Antigen-Directed Induction Therapy for Newly Diagnosed Patients With B-Cell Precursor Acute Lymphoblastic Leukemia and Lymphoma
Brief Title: Therapy for Newly Diagnosed Patients With B-Cell Precursor Acute Lymphoblastic Leukemia and Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Pfizer (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJALL23H; NCI-2024-06013 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Newly Diagnosed; Antigen-directed therapies; Induction therapy; Children; Young Adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; Calcium Dobesilate; Vincristine; Inotuzumab Ozogamicin; blinatumomab; Dasatinib; Methotrexate; Hydrocortisone; Cytarabine; Cyclophosphamide; Mercaptopurine; calaspargase pegol; Daunorubicin; Thioguanine

STUDY DESIGN:
Intervention Model Description: This study utilizes a single arm phase II design enrolling eligible participants with newly diagnosed B-cell precursor acute lymphoblastic leukemia and lymphoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SJALL23H Treated Patients (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Induction: Dexamethasone, Vincristine, Inotuzumab, Blinatumomab, Cyclophosphamide, Dasatinib, IT MHA.
  Early Post Induction: Cyclophosphamide, Cytarabine, Inotuzumab, Methotrexate, IT MHA, Dasatinib, Blinatumomab, 6-mercaptopurine, Dexamethasone, Vincristine, Daunorubicin, Calaspargase.
  Maintenance: Dexamethasone, Vincristine, Methotrexate, 6-mercaptopurine, Thioguanine, Dasatinib, IT MHA.
  Interventions: Drug: Dexamethasone; Drug: Vincristine; Drug: Inotuzumab; Drug: Blinatumomab; Drug: Dasatinib; Procedure: IT MHA; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Methotrexate; Drug: 6-Mercaptopurine; Drug: Calaspargase; Drug: Daunorubicin; Drug: Thioguanine

INTERVENTIONS:
Drug: Dexamethasone — Given orally (PO) or intravenously (IV).
  Other Names: Decadron; Hexadrol®
Drug: Vincristine — Given IV.
  Other Names: Vincristine Sulfate; Oncovin
Drug: Inotuzumab — Given IV.
  Other Names: Inotuzumab ozogamicin; BESPONSA®
Drug: Blinatumomab — Given IV.
  Other Names: BLINCYTO®
Drug: Dasatinib — Given PO.
  Other Names: Sprycel®
Procedure: IT MHA — Given Intrathecal (IT), Age adjusted.
  Other Names: Intrathecal triple therapy (methotrexate + hydrocortisone + cytarabine)
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan®
Drug: Cytarabine — Given IV or IT.
  Other Names: Cytosine arabinoside; Ara-C
Drug: Methotrexate — Given IT, IV, PO or intramuscular (IM).
  Other Names: MTX; Trexall®
Drug: 6-Mercaptopurine — Given PO.
  Other Names: Mercaptopurine; 6-MP
Drug: Calaspargase — Given IV.
  Other Names: ASPARLAS
Drug: Daunorubicin — Given IV.
  Other Names: Daunomycin
Drug: Thioguanine — Given PO (participants intolerant to mercaptopurine).
  Other Names: 6-thioguanine; Tabloid®

SUMMARY:
This is a Phase II clinical trial testing the use of two antigen-directed therapies, inotuzumab and blinatumomab, as part of induction therapy for children and young adults with newly diagnosed B-cell precursor acute lymphoblastic leukemia and lymphoma.

Primary Objective

* To assess if the flow-cytometry assessed MRD-negative remission rate following an immunotherapy-based Induction in NCI-high risk patients without favorable genetic features is higher than the results of similar patients treated on AALL1131.

Secondary Objectives

* To compare flow-cytometry assessed MRD-negative rates at the end of Induction for patients treated with this therapy compared to similar patients treated on TOT17.
* To compare the rate of significant toxicities in patients treated with this therapy to those treated with standard-risk therapy on TOT17.
* To assess the event free and overall survival of patients treated with this therapy.

DETAILED DESCRIPTION:
This study utilizes a single arm phase II design. Treatment will consist of 3 main phases: Induction, early post induction [including Consolidation, Blinatumomab 1, High-Dose Methotrexate, Reinduction, Interim, Reconsolidation, and Blinatumomab 2], and Maintenance.

Induction:

* Induction includes 7 days of therapy on the INITIALL classification protocol (NCT06289673) as well as 5 further weeks of treatment on this trial. Treatment includes 15 days of oral (PO) or intravenous (IV) dexamethasone, 3 weekly doses of vincristine IV, and 2 doses of inotuzumab IV on Days 2 and 8. Patients will then receive blinatumomab IV from Days 9-36. Dasatinib PO will be added beginning on Day 12 for patients with an ABL-class fusion including patients with Ph+ ALL. These patients will also receive dasatinib in all subsequent cycles of therapy. Intrathecal (IT) MHA will be given. Patients will have a week without chemotherapy at the end of Induction, although patients with Induction failure (MRD ≥5% disease) will proceed directly to consolidation. Patients unable to receive inotuzumab by day 3 receive cyclophosphamide IV on days 3-4.

Early Post Induction:

* Consolidation will be given following completion of Remission Induction Therapy. Patients receive cyclophosphamide intravenous (IV), cytarabine IV, inotuzumab IV, intrathecal (IT) MHA, and dasatinib PO for patients with ABL-class fusion. Patients will have a week without chemotherapy at the end of Consolidation.
* Blinatumomab 1 will be given with IT MHA for four weeks to all patients after recovery from Consolidation.
* High-dose Methotrexate will be given IV every two weeks for four cycles. Patients will also receive an IT MHA with each of the 2 week cycles and will take oral mercaptopurine continuously if tolerated.
* Reinduction will consist of dexamethasone for 7 days in the first and third week, 3 weekly doses of vincristine IV, 1 dose of daunorubicin IV, 1 dose of calaspargase IV, intrathecal (IT) MHA one dose, and dasatinib PO daily (for patients with ABL-class fusion).
* Interim includes mercaptopurine po daily for 6 weeks, dexamethasone for 1 week (5 days), daunorubicin and vincristine IV on day 1 of weeks 2 and 5, calaspargase IV on day 1 of weeks 1 and 4, IT MHA on day 1 of week 4 and dasatinib po daily for 6 weeks (for patients with ABL-class fusion). Patients will have a week without chemotherapy at the end of Interim Therapy. Patients with Down syndrome will not receive daunorubicin during this phase.
* Reconsolidation will repeat therapy given in Consolidation but replace the investigational inotuzumab with traditional mercaptopurine.
* Blinatumomab 2 will be given for four weeks to patients without clonal IgH rearrangements, those with end of Induction MRD, those in whom next-generation based sequencing MRD is unavailable, patients who did not receive blinatumomab during induction, or patients with Down syndrome after Reconsolidation.

Maintenance therapy follows Reconsolidation or Blinatumomab 2 (for those patients receiving this therapy) and includes 8 pulses of dexamethasone and vincristine given every 4 weeks, weekly methotrexate, daily mercaptopurine, intrathecal therapy, and dasatinib (for patients with ABL-class fusions). Maintenance therapy lasts a total of 80 weeks.

Duration of therapy is approximately 2¼ years. Follow-up is recommended until the patient is in remission for 10 years and is at least 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on INITIALL.
* Age 1-18.99 years at the time of enrollment on INITIALL.
* B-Acute lymphoblastic leukemia or lymphoblastic lymphoma.
* No prior chemotherapy excluding therapy given on or allowed by INITIALL.
* NCI high-risk (age 10 years or greater or presenting WBC count ≥50,000 cells/microL) or NCI standard-risk and a HR clinical feature as listed below:

  * CNS3 disease (≥5 WBC/microL CSF with blasts present)
  * Testicular involvement of leukemia
  * Steroid pretreatment defined as >24 hours of therapy in the 14 days prior to enrollment on INITIALL if a preceding WBC to define NCI risk is unavailable
* For lymphoblastic lymphoma, Stage 3-4 disease OR Stage 1-2 disease in patient ages ≥10 years OR HR clinical feature as defined above.
* Adequate liver function defined as:

  * Total bilirubin ≤ 1.5x the upper limit of normal for age and alanine transaminase (ALT) ≤ 5x the upper limit of normal for age. Patients with an elevated total bilirubin due to hemolysis are eligible if they have a direct bilirubin <1.5x the upper limit of normal.
* Adequate renal function defined as:

  * Calculated glomerular filtration rate (GFR) ≥ 50 mL/min/1.73m^2 using the Bedside Schwartz equation OR creatinine below or equal to the maximum defined below:

    * Age: 1 to <2 years; maximum serum creatinine (mg/dL): 0.6 (male and female)
    * Age: 2 to <6 years; maximum serum creatinine (mg/dL): 0.8 (male and female)
    * Age: 6 to <10 years; maximum serum creatinine (mg/dL): 1.0 (male and female)
    * Age: 10 to <13 years; maximum serum creatinine (mg/dL): 1.2 (male and female)
    * Age: 13 to <16 years; maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
    * Age: ≥16 years; maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)
* Eligibility for inclusion post-induction requires meeting the first 4 Inclusion criteria above AND:

  * Treatment on SJALL23H for Induction OR
  * Lymphoblastic lymphoma, initially treated on an SJALL protocol OR standard (non-protocol) therapy, without a complete response at the end of induction OR
  * NCI-SR ALL at diagnosis and treated with an SJALL protocol OR standard (non-protocol) therapy who have

    * Slow response to therapy (≥0.1% MRD at end of induction for patients with hyperdiploid ALL or ≥0.01% MRD at end of induction for others with ALL) OR
    * HR genetics as defined in the protocol.
    * These patients may receive no more than 2 weeks of post-induction therapy and should be transitioned to SJALL23H post-induction as soon as the qualifying genetic or MRD result is available.

Exclusion Criteria:

* Presence of ETV6::RUNX1 fusion unless also having a HR clinical feature OR slow response to induction therapy.
* History or presence of clinically relevant central nervous system (CNS) pathology or event such as epilepsy, childhood or adult non-febrile seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. History of simple febrile seizure during childhood and presence of CNS leukemia at diagnosis are not exclusions to participation.
* Active uncontrolled infection.
* Current active autoimmune disease or history of autoimmune disease with the potential for CNS involvement.
* History of venoocclusive disease/ sinusoidal obstructive syndrome.
* Unstable cardiac disease including QTc >500msec.
* Inability or unwillingness to give informed consent/ assent as applicable.
* Pregnant or lactating.
* For patients of reproductive potential, unwillingness to use effective contraception for the duration of protocol therapy.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
End of induction minimal residual disease negative remission | On treatment to end of induction, approximately 29 days
  Flow cytometry (preferred) or next generation sequencing measurement of bone marrow with <0.01% leukemia with resolution of extramedullary disease at the end of induction (approximately day 29) and will be analyzed within 6 months of the last participant reaching the timepoint.

SECONDARY OUTCOMES:
Comparison of MRD-negative rates to those on Total 17 | On treatment to end of induction, approximately 29 days
  Flow cytometry (preferred) or next generation sequencing measurement of bone marrow with <0.01% leukemia with resolution of extramedullary disease will be compared between patients enrolled on this trial and patients with similar clinical features (age, WBC at diagnosis, CNS status, testicular involvement) enrolled on Total 17(NCT03117751).
Compare significant toxicities experienced to those on Total 17 | On treatment to end of reconsolidation, approximately 56 days.
  We will compare CTCAE version 5 clinically significant, non-hematological grade 3 or any non-hematological grade 4-5 toxicities. This comparison will encompass 3 periods: induction/ consolidation, reinduction, and reconsolidation.
Event free survival (EFS) | 3.5 years after enrollment.
  Kaplan-Meier estimates of the survival functions for event-free survival (EFS) will be calculated along with standard error. For EFS, death due to any cause, any relapse, consolidation failure, and second malignancy are considered as failure; patients remaining failure-free at the last follow up are censored.
Overall survival (OS) | 3.5 years after enrollment.
  Kaplan-Meier estimates of the survival functions for overall survival (OS) will be calculated along with standard error. For OS, only death due to any cause is considered as failure and patients still alive at the last follow up are censored.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Karol, MD, MSCI, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Saint Francis Children's Hospital, Tulsa, Oklahoma
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols